CLINICAL TRIAL: NCT03745755
Title: Derivation of a Clinical Decision Rule for Emergency Department Head CT Scanning in Seniors Who Have Fallen (the Falls Multicentre Study)
Brief Title: Derivation of a Clinical Decision Rule for Emergency Department Head CT Scanning in Seniors Who Have Fallen
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Falls_MC_5304
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Fall; Intracranial Bleed
Keywords: elderly; clinical decision rule; emergency department; CT scan; bleeding
MeSH Terms: conditions — Intracranial Hemorrhages; Emergencies; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Falls are the leading cause of traumatic death in the elderly with head injury causing half of these deaths. Each year, one in three adults over the age of 65 (seniors) fall, and half of these seniors seek treatment at a hospital emergency department (ED). There is a major evidence gap in the study of brain injury diagnosis in seniors, which is problematic for emergency physicians since the number of fall-associated head injuries is rising. ED diagnostic tools for risk stratification of these patients do not exist. The investigators will derive a novel ED clinical decision rule for detecting traumatic intracranial bleeding which will standardize the approach to head CT scans. Once validated, the investigators will optimize patient care by ensuring that intracranial bleeding is identified early. By reducing the use of head CT, this decision rule will lead to health care savings and streamlined, patient-centered ED care.

DETAILED DESCRIPTION:
This study is designed to develop a unique clinical decision rule for ED physicians evaluating senior patients who have fallen. Clinical decision rules are a common method for standardizing diagnostic decision-making and minimizing misdiagnosis in the ED. Each patient will be assessed at their index ED visit by an emergency physician who will record history and examination findings. The primary outcome will be clinically important intracranial bleeding diagnosed with 42 days. Patients who return to the ED within 42 days with new confusion, headache, loss of balance, repeat falls, change in behaviour, reduced Glasgow Coma Scale score or other neurological symptoms will also undergo head CT. All intracranial bleeding events will be adjudicated independently.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years old
* Fall within 48 hours of emergency department visit (regardless of presenting complaint)

Exclusion Criteria:

* Repeat event/visit (already enrolled in the study)
* Transferred from another hospital
* Lives outside of hospital catchment area
* Major trauma (e.g. fall from steps, fall from height, motor vehicle accident, struck by a vehicle, recreational accident)
* Left emergency department prior to completion of assessment (left against medical advice)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: ED patients aged over 65 years who present to the ED within 48 hours of having a fall. Eligibility is determined by having fallen on level ground (either inside or outside), off a chair or toilet seat or off a bed.
  Patients are included regardless of whether they hit their head.
Sampling Method: Non-Probability Sample
Enrollment: 4308 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Clinically important intracranial bleeding | Within 42 days of the index emergency department presentation.
  Number of patients with bleeding within the cranial vault (including subdural, intracerebral, intraventricular, subarachnoid, epidural blood and cerebral contusion) which requires medical or surgical treatment.

SECONDARY OUTCOMES:
Neurosurgical intervention | Within 90 days
  Number of patients with intracranial bleeding who undergo neurosurgical intervention.
Intensive care admission | Within 90 days
  Number of patients with intracranial bleeding who are admitted to the intensive care unit.
Hospital length of stay | Within 90 days
  Duration of hospitalization among patients with intracranial bleeding.
In-hospital death | Within 90 days
  Number of patients with intracranial bleeding who die in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin de Wit, MD, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] de Wit K, Mercuri M, Clayton N, Mercier E, Morris J, Jeanmonod R, Eagles D, Varner C, Barbic D, Buchanan IM, Ali M, Kagoma YK, Shoamanesh A, Engels P, Sharma S, Worster A, McLeod S, Emond M, Stiell I, Papaioannou A, Parpia S; Network of Canadian Emergency Researchers. Derivation of the Falls Decision Rule to exclude intracranial bleeding without head CT in older adults who have fallen. CMAJ. 2023 Dec 3;195(47):E1614-E1621. doi: 10.1503/cmaj.230634. PMID 38049159
- [Derived] de Wit K, Mercuri M, Clayton N, Worster A, Mercier E, Emond M, Varner C, McLeod SL, Eagles D, Stiell I, Barbic D, Morris J, Jeanmonod R, Kagoma Y, Shoamanesh A, Engels PT, Sharma S, Kearon C, Papaioannou A, Parpia S; Network of Canadian Emergency Researchers. Which older emergency patients are at risk of intracranial bleeding after a fall? A protocol to derive a clinical decision rule for the emergency department. BMJ Open. 2021 Jul 2;11(7):e044800. doi: 10.1136/bmjopen-2020-044800. PMID 34215600